CLINICAL TRIAL: NCT02269215
Title: A Single Blind, Placebo-controlled, Parallel-group, Single Increasing Dose Tolerance Study in Healthy Young Male Volunteers After Intravenous Administration of BIII 890 CL as Loading Dose (Dosage: 12.5, 25, 50 mg/h, Infusion Time 1 hr; 50 mg/h, Infusion Time 2 Hrs) Followed by Maintenance Dose (Dosage: 6.25, 12.5, 25 mg/h, Infusion Time 5 Hrs; 30 mg/h, Infusion Time 4 Hrs) and in Healthy Elderly Male and Female Volunteers After Intravenous Administration of BIII 890 CL as Loading Dose (Dosage: 50 mg/h, Infusion Time 1 hr) Followed by Maintenance Dose (Dosage: 25 mg/h, Infusion Time 5 Hrs)
Brief Title: Single Increasing Doses of BIII 890 CL in Healthy Young Male Volunteers and in Healthy Elderly Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 599.2
Record Dates: First submitted 2014-10-20; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — BIII 890 CL

ARMS (2):
- BIII 890 CL single rising dose (Experimental)
  Interventions: Drug: BIII 890 CL
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIII 890 CL
  Arms: BIII 890 CL single rising dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
Safety, tolerability and pharmacokinetics of BIII 890

ELIGIBILITY:
Inclusion Criteria:

* Participants in the study should be healthy males, range from 21 to 50 years of age and be within +- 20% of their normal weight (Broca-Index) and healthy elderly males and females, > 60 years of age and be within +-25 % of their normal weight (Broca-Index)
* In accordance with good clinical practice (GCP) and the local legislation all volunteers will have given their written informed consent prior to admission to the study

Exclusion Criteria:

* Volunteers were excluded from the study if the results of the medical examination, laboratory tests or ECG recordings are judged by the investigator to differ significantly from normal clinical values
* Volunteers with known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Volunteers with diseases of the central nervous system (such as epilepsy), central nervous system (CNS) trauma in their medical history or with psychiatric disorders or neurological disorders
* Volunteers with known history of relevant orthostatic hypotension, fainting spells or blackouts
* Volunteers with chronic or relevant acute infections
* Volunteers with history of allergy/hypersensitivity (including drug allergy) which was deemed relevant to the trial as, judged by the investigator
* Volunteers who had taken a drug with a long half-life (≥ 24 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study
* Volunteers who received any other drugs which could influence the results of the trial during the week prior to the start of the study
* Volunteers who participated in another study with an investigational drug within the last two months preceding this study
* Volunteers who smoke (> 10 cigarettes or 3 cigars or 3 pipes/day)
* Volunteers who were not able to refrain from smoking on study days
* Volunteers who drunk more than 60 g of alcohol per day
* Volunteers who were dependent on drugs
* Volunteers who participated in excessive physical activities (e.g. competitive sports) during the last week before the study
* Volunteers who donated blood within the last 4 weeks (≥ 100 mL)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2000-01; Primary Completion 2000-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with clinically relevant changes in vital signs | Pre-dose, up to 8 days after drug administration
  blood pressure, pulse rate, respiratory rate, body temperature
Number of subjects with clinically relevant changes in 12-lead ECG | Pre-dose, up to 8 days after drug administration
Number of subjects with clinically relevant changes in laboratory parameters | Pre-dose, up to 8 days after drug administration
  including coagulation parameters
Number of subjects with adverse events | Up to 8 days after drug administration

SECONDARY OUTCOMES:
Maximum measured concentration of the analyte in plasma (Cmax) | up to 32 hours after start of drug administration
Time from dosing to the maximum concentration of the analyte in plasma over a uniform dosing interval λz (tmax) | up to 32 hours after start of drug administration
Apparent terminal half-life of the analyte in plasma (t1/2) | up to 32 hours after start of drug administration
Area under the concentration-time curve of the analyte in plasma (AUC) | up to 32 hours after start of drug administration
Mean residence time (MRT) | up to 32 hours after start of drug administration
Plasma clearance (CL) | up to 32 hours after start of drug administration
Volume of distribution (V) | up to 32 hours after start of drug administration
Amount of parent drug excreted into urine (Ae) | up to 32 hours after start of drug administration